CLINICAL TRIAL: NCT05713201
Title: Percutaneous Coronary Interventions of the Aneurysmatic and Ectasic Right Coronary Artery in the Acute Setting: Management and Immediate- and Long-Term Outcomes The RIGHT-MARE Study
Brief Title: Outcomes After PCI of the Aneurysmatic Right Coronary Artery
Acronym: RIGHT-MARE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Principal investigator, San Luigi Gonzaga Hospital
Other Study IDs: 001-2022
Record Dates: First submitted 2023-01-23; First posted 2023-02-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Coronary Disease; Coronary Artery Ectasia; Right Coronary Artery Occlusion; Right Coronary Artery Stenosis; STEMI
Keywords: PCI; Acute Coronary Syndrome; Aneurysmatic Right Coronary Artery
MeSH Terms: conditions — Coronary Disease; Coronary Aneurysm; ST Elevation Myocardial Infarction; Acute Coronary Syndrome | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index PCI: Patients with an aneurysmatic right coronary artery undergoing index PCI in the acute setting.
  Interventions: Procedure: Percutaneous Coronary Intervention
- Staged PCI: Patients with an aneurysmatic right coronary artery undergoing staged PCI in the acute setting.
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Treatment of coronary stenoses with a drug-eluting stent or balloon

SUMMARY:
This study aims to evaluate procedural and clinical outcomes of acute coronay syndrome (ACS) patients with aneurysmatic culprit right coronary artery (RCA).

DETAILED DESCRIPTION:
The investigators sought differences in procedural (slow-flow, no-reflow, distal embolisation,Thrombolysis in Myocardial Infarction final flow (TIMI) etc.) and in immediate and long-term clinical outcomes between several subgroups such as index vs staged percutaneous coronary intervention (PCI), premedication vs none, use of IIb/IIIa inhibitors vs none, bare metal stent (BMS) vs drug eluting stent (DES), ultrathin DES vs thick DES, durable polymer vs bioresorbable or free polymer etc.

The investigators also want to investigate the efficacy of different technical manoeuvres involved in resolving high thrombotic burden before stent deployment, such as thrombus aspiration, dilatation, intracoronary infusion of adenosine or thrombolytic agents, direct stenting etc.). Long-term follow-up includes target vessel failure (Cardiac Death, target vessel MI, clinically-driven target vessel revascularisation), define or probable stent thrombosis, target vessel revascularisation for ACS, clinically driven target vessel revascularisation and intrastent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ACS of the aneurysmatic or ectasic RCA
* Patient with at least 6 months clinical or angiographic follow-up
* Patients with accurate procedural and clinical records (particularly use of drugs before, during and after procedure, according to RCA PCI procedure (index or staged).

Exclusion Criteria:

* Elective aneurysmatic or ectasic RCA PCI
* Patient with lack of accurate procedural and clinical data
* Patient with lack of clinical or angiographic follow up

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with aneurysmatic or ectatic right coronary artery disease in the acute setting following PCI.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | Procedural (from the start to the end of the procedure)
  Defined as final TIMI flow > 3 (TIMI 0: absence of any integrate flow beyond the coronary occlusion; TIMI 1: faint antegrade flow beyond the coronary occlusion with incomplete filling of the distal coronary bed; TIMI 2: delayed flow beyond the coronary occlusion with complete filling of the distal coronary bed; TIMI 3: normal flow with complete filling of the distal coronary bed)

SECONDARY OUTCOMES:
Target Lesion Failure | 12 moths
  Combination of cardiac death, target vessel MI and clinically target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (8):
- Italy (6):
  - Ospedale Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Brotzu, Cagliari
  - Policlinico Universitario G.Rodolico, Catania
  - Azienda Ospedaliera Universitaria Gaetano Martino, Messina
  - Ospedale Auxologico San Luca, Milan
  - Interventional Unit, San Luigi Gonzaga University Hospital, Orbassano, and Rivoli Hospital, Turin, Italy, Turin
- Spain (2):
  - Ospedale Universitario Marqués de Valdecilla, Santander, Satander
  - Hospital Clinico San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No